CLINICAL TRIAL: NCT06280807
Title: OBServation of Environment and ReproductiVe Endocrine Effects Study (OBSERVE Study)
Brief Title: Observation of Environment and Reproductive-Endocrine Effects
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001617; 001617-E
Record Dates: First submitted 2024-02-24; First posted 2024-02-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-19

CONDITIONS: Hypogonadism; Hypergonadism; Precocious Puberty; Late Puberty; Amenorrhea
Keywords: Endocrine; Reproductive Disorders; Hypothalamic-Pituitary-Gonadal Endocrine Axis
MeSH Terms: conditions — Hypogonadism; Puberty, Precocious; Amenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Androgen Excess States: Polycystic Ovary Syndrome (PCOS);Women who meet criteria for PCOS based on NIH/ Rotterdam or other clinical criteria
- Congenital Adrenal Hyperplasia / Hyperandrogenism: Women who exhibit evidence of hyperandrogenism not related to Polycystic Ovarian Syndrome (PCOS); Nonclassic Congenital Adrenal Hyperplasia, Extreme hyperinsulism, Idiopathic etc.
- Exhibiting signs of a diagnosis of hypogonadism: for example: Bosma arrhinia microphthalmia syndrome (BAMS)
- Hypogonadism / Infertility: Isolated hypogonadotropic hypogonadism
- Hypothalamic Amenorrhea (HA) (female) Functional Hypogonadism (male): Participants who experience secondary or primary amenorrhea, or male hypogonadism, in the setting of negative energy balance such dieting, eating disorders or exercise training
- Miscellaneous: Reproductive disorders not related to the above categories. (e.g., secondary to endocrine dysfunction, thyroid disorders, Cushing syndrome, pharmacotherapy, etc.)
- Precocious or Delayed Puberty: Participants who display clinical evidence of delayed or precocious puberty based on standard criteria.
- Premature Ovarian InsufficiencyPerimenopause or post-menopausal states: Women who attain menopause before age 40 years (or as defined by clinical criteria). Perimenopausal women are those typically above age 40 years and experience secondary amenorrhea/ oligomenorrhea.
- Weight *Overweight/Underweight: BMI below or above reference standard (Adult Reference: Asians/ Asian Americans- 18.5-22.9 kg/m2; Other races- 18.5-24.9 kg/m2*Participants may simultaneously belong to cohort of weight and any other cohort.

SUMMARY:
Background:

Endocrine disorders occur when the glands that make hormones do not work properly. Hormones levels that are too high or too low can cause problems such as late or early puberty, irregular periods, and infertility. Environmental factors - including pollution; chemical exposure at home and work; foods; medicines; and sleep habits - may cause problems with the endocrine and reproductive systems.

Objective:

To learn how environmental factors may affect the endocrine and reproductive systems.

Eligibility:

Males or females, referring to sex assigned at birth, aged 8 years and older; they must have hypogonadism, infertility, or other reproductive disorders.

Design:

Adult participants will have 4 to 5 visits in 5 years. Children may have up to 12 visits; they may remain in the study up to the age of 23. Most visits will be less than 3 hours.

Participants will be screened. They will have a physical exam. They will have blood and urine tests. They will complete questionnaires; they will answer questions about their diet, health, and other topics. Some may be referred for additional tests, such as imaging scans and semen analysis.

Specific tests conducted during study visits will vary, depending on the participant s diagnosis. In addition to repeated blood and urine tests, these may include:

Body composition measure: Participants will sit in a pod-shaped machine for about 6 minutes. The machines measures the air inside the capsule to record body fat and breathing volume.

Resting energy expenditure test: Participants will lie down with a clear dome placed over their head. They will breathe quietly for 30 minutes. This test measures the number of calories their body burns at rest.

...

DETAILED DESCRIPTION:
Study Description:

This study will investigate the relationship between environment, lifestyle, and reproductive function. This will include the study of these factors at enrollment and in response to clinical care for the underlying condition. This study will prospectively follow participants with endocrine reproductive disorders and collect data secondary to clinical care and data regarding internal and external environmental exposures. We hypothesize that dysregulated environment is associated with reproductive and endocrine dysfunction and the clinical phenotype may evolve in response to treatment of the dysfunction. To study the hypothesis that external and internal environmental factors are associated with reproductive and endocrine dysfunction.

Objectives:

* To study the hypothesis that external and internal environmental factors are associated with reproductive and endocrine dysfunction
* To generate hypothesis for future studies investigating the impact of environment on human health

Endpoints:

Since this is an exploratory and hypothesis generating study there are no pre-defined endpoints of this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, referring to sex assigned at birth (cis gender)
2. Age > 8 years and weight >= 12 kg
3. A diagnosis of hypogonadism, infertility or other reproductive dysfunction

   Some specific diagnoses (as defined in standard guidelines) will include:
   * Male or female hypogonadism

     * Obesity/metabolic syndrome related to hypogonadism.
     * Other reproductive dysfunction (e.g., secondary to endocrine dysfunction, thyroid disorders, Cushing syndrome, pharmacotherapy, etc.)
     * Premature Ovarian Insufficiency
     * Isolated hypogonadotropic hypogonadism
   * Polycystic Ovarian Syndrome
   * Delayed Puberty
   * Precocious puberty
   * Perimenopause and post-menopausal states
   * Androgen Excess States (Nonclassic Congenital Adrenal Hyperplasia, Extreme hyperinsulism, Idiopathic etc.)

   or

   -Exhibiting signs of a diagnosis of hypogonadism, e.g., Bosma arrhinia microphthalmia syndrome (BAMS)
4. Ability of participant, legal guardian, or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. A diagnosis of a serious medical disorder such as malignancy or heart disease will be grounds for exclusion at the discretion of the PI or AI.
2. Inability to follow up with the research study and/or perform study procedures, at the discretion of the PI or AI.
3. Pregnant participants, less than 18 years of age, for their safety, since there is not a trained doctor on the study to give proper medical care to pregnant individuals less than 18 years of age.

Individuals who do not meet the criteria for participation in this study (screen failure) because of an acute, reversible or transient medical reason may be rescreened upon reversal, improvement or stabilization of their clinical status. Participants who develop an acute, reversible or transient medical condition during the study may return upon reversal, improvement or stabilization of their clinical status.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric (between the ages of 8 and 18), cisgender male and females, from the communities and surrounding areas of Durham, Chapel Hill and Raleigh in NC; and Bethesda, MD.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2039-03-28 (Estimated); Study Completion 2039-03-31 (Estimated)

PRIMARY OUTCOMES:
Investigate the relationship between environment, lifestyle, and reproductive neuroendocrinology. | at baseline and after clinical care for the underlying condition
  We will analyze the correlation between internal exposures, and the longitudinal evolution of endocrine disorders. For instance, changes in PSQI (sleep) and DSM-5 (mood) questionnaire scores, research analytes and hormone metrics with treatment.

SECONDARY OUTCOMES:
the relationship between nutrition, diet and reproduction | at baseline and after clinical care for the underlying condition
  We will analyze the correlation between external exposures, and the longitudinal evolution of endocrine disorders. For instance, we will assess for changes in (stress), eating disorders and exposome information (derived from co-enrollment in the PEGS study) before and after treatment.
the impact of stress on reproductive dysfunction | at baseline and after clinical care for the underlying condition
  We will analyze the correlation between external exposures, and the longitudinal evolution of endocrine disorders. For instance, we will assess for changes in (stress), eating disorders and exposome information (derived from co-enrollment in the PEGS study) before and after treatment.
the influence of behavioral and psychological factors on reproductive function | at baseline and after clinical care for the underlying condition
  We will analyze the correlation between external exposures, and the longitudinal evolution of endocrine disorders. For instance, we will assess for changes in (stress), eating disorders and exposome information (derived from co-enrollment in the PEGS study) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie D Shaw, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated and summarized data will be made available as part of associated publication, using NIH-Supported Data Sharing Resources (nlm.nih.gov/NIHbmic/generalist_repositories.html )@@@Aggregated summary and statistical analysis will be publicly available. All the patient-level data will require controlled access.@@@Outside investigators may apply for research collaborations related to the original research questions, that will be IRB approved for use and a data transfer agreement will be signed, and coded, deidentified data will be provided with a data dictionary. For studies unrelated to the original research, only deidentified data can be provided and only when subjects consented to future research.@@@Summary clinical response and adverse event data will be placed in clinicaltrials.gov one year after the final subject has completed the primary endpoint. @@@
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available with the scientific publication upon reasonable request. In some cases, especially per journal policy and as appropriate, we will deposit deidentified data.
Access Criteria: Aggregated summary and statistical analysis will be publicly available. All the patient-level data will require controlled access.

REFERENCES:
- [Background] Moran LJ, Hutchison SK, Norman RJ, Teede HJ. Lifestyle changes in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD007506. doi: 10.1002/14651858.CD007506.pub3. PMID 21735412
- [Background] Sharma R, Biedenharn KR, Fedor JM, Agarwal A. Lifestyle factors and reproductive health: taking control of your fertility. Reprod Biol Endocrinol. 2013 Jul 16;11:66. doi: 10.1186/1477-7827-11-66. PMID 23870423
- [Background] Roychoudhury S, Chakraborty S, Choudhury AP, Das A, Jha NK, Slama P, Nath M, Massanyi P, Ruokolainen J, Kesari KK. Environmental Factors-Induced Oxidative Stress: Hormonal and Molecular Pathway Disruptions in Hypogonadism and Erectile Dysfunction. Antioxidants (Basel). 2021 May 24;10(6):837. doi: 10.3390/antiox10060837. PMID 34073826
- [Background] Corona G, Rastrelli G, Morelli A, Sarchielli E, Cipriani S, Vignozzi L, Maggi M. Treatment of Functional Hypogonadism Besides Pharmacological Substitution. World J Mens Health. 2020 Jul;38(3):256-270. doi: 10.5534/wjmh.190061. Epub 2019 Aug 29. PMID 31496147
- [Background] Gravholt CH, Chang S, Wallentin M, Fedder J, Moore P, Skakkebaek A. Klinefelter Syndrome: Integrating Genetics, Neuropsychology, and Endocrinology. Endocr Rev. 2018 Aug 1;39(4):389-423. doi: 10.1210/er.2017-00212. PMID 29438472
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001617-E.html